CLINICAL TRIAL: NCT00363636
Title: A Phase III, Randomized, Double-Blind Study of Galiximab in Combination With Rituximab Compared With Rituximab in Combination With Placebo for the Treatment of Subjects With Relapsed or Refractory, Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study of Galiximab + Rituximab Versus Rituximab + Placebo in Follicular Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment challenges due to changes in standards of care resulted in premature termination. No safety or efficacy events factored into this action.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114-NH-301
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2011-03

CONDITIONS: Lymphoma, Non-Hodgkin's
Keywords: relapsed; NHL; pharmacokinetics; antibody; safety; galiximab; efficacy; rituximab; refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — galiximab; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Galiximab in combination with rituximab
- 2 (Active Comparator)
  Interventions: Drug: Rituximab in combination with placebo

INTERVENTIONS:
Drug: Galiximab in combination with rituximab — Galiximab (500mg/m2 IV) in combination with Rituximab (375 mg/m2 IV), weekly x 4
  Arms: 1
Drug: Rituximab in combination with placebo — Rituximab (375 mg/m2 IV) in combination with placebo, weekly x 4
  Arms: 2

SUMMARY:
This is a Phase III, multicenter, global, clinical study of an investigational drug called galiximab in combination with an approved drug called rituximab in subjects with follicular NHL.

The purpose of the study is to compare the clinical benefit of galiximab when given in combination with rituximab as compared with rituximab alone (given with placebo) in subjects with follicular NHL. Safety and pharmacokinetics (PK) of galiximab and rituximab will also be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

Key Inclusion Criteria:

* Aged >= 18 years old at the time of informed consent.
* Histologically confirmed follicular Grade 1-3a NHL.
* Relapsed or progressive disease after at least 1 prior chemotherapy requiring treatment.
* Bidimensionally measurable disease with at least 1 lesion >= 2.0 cm in a single dimension.
* Acceptable hematologic, hepatic, and renal function parameters.
* Recovered fully from any significant toxicity associated with prior surgery, radiation treatments, chemotherapy, biological therapy, autologous bone marrow or stem cell transplant, or investigational drugs.

Key Exclusion Criteria:

* Follicular lymphoma Grade 3b.
* Rituximab refractory or refractory to anti-CD20 radioimmunotherapy (no response to prior rituximab or prior rituximab-containing regimen, or a response with a TTP of less than 6 months).
* Cancer radiotherapy, biological therapy, or chemotherapy within 3 weeks prior to Study Day 1 (6 weeks if nitrosourea or mitomycin C).
* Prior lymphoma vaccine therapy within 12 months prior to Study Day 1.
* Prior antibody therapy for lymphoma (including radioimmunotherapy) within 6 months prior to Study Day 1.
* Autologous bone marrow or stem cell transplant within 6 months prior to Study Day 1.
* Prior allogeneic transplant.
* Transfusion-dependent subjects.
* Another primary malignancy requiring active treatment (except hormonal therapy).
* Serious nonmalignant disease (e.g., congestive heart failure, hydronephrosis); active uncontrolled bacterial, viral, or fungal infections; or other conditions, which would compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
* New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to Study Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To assess efficacy as measured by progression free survival (PFS), and determine whether rituximab plus galiximab compared to rituximab plus placebo may extend PFS. | The duration of this study is approx 4 years

SECONDARY OUTCOMES:
Secondary efficacy measures include: event-free survival, time to progression, duration of response, complete response rate, and overall survival. | The duration of this study is approx 4 years
Safety measures include: adverse event rates, clinical laboratory results, development of anti-galiximab and human anti-chimeric antibodies. | The duration of this study is approx 4 years
Pharmacokinetics | The duration of this study is approx 4 years
Quality of Life using both the Functional Assessment of Cancer Therapy-Lymphoma (FACT-lym) and the EQ-5D (EuroQoL) instruments | The duration of this study is approx 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen